CLINICAL TRIAL: NCT00526604
Title: A Study on the Effect of Employment Follow-up on Return to Work in Sick Listed Patients With Low Back Pain
Brief Title: Work Related Rehabilitation in Patients With Low Back Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped, as the another multicentre-RCT on the same patients started.
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Anne Keller, Ulleval University Hospital, 0407 Oslo, Norway
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Work and LBP
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-12

CONDITIONS: Low Back Pain
Keywords: return to work; low back pain; work related rehabilitation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Active Comparator): The control group will have an clinical examination and exercise and then return to general practitioner, which will take decision about sick leave or return to work.
  Interventions: Behavioral: work related rehabilitation

INTERVENTIONS:
Behavioral: work related rehabilitation — The workplace intervention includes two steps:
  Evaluations of the work site: The occupational ergonomists task is to identify conditions at the work site, as for instance ergonomic, work demand and relations to the employer and colleagues.
  Therapeutic Return to work: The occupational ergonomists will organize contacts and meetings between the employer and the patients and make a schedule for return to work. The therapeutic return-to-work-process will take place at the work place, with progressively more days at work and progressively increasing tasks.

SUMMARY:
Low back pain is a usual conditions in the western countries and several treatments available for patients with "non-specific low back pain". According to the European guidelines are exercise and cognitive intervention effective on pain and function(www.backpaineurope.org), but it have no documented effect on return to work. In addition, there is no documentation that treatments which focus on a single treatment, is effective with regard to return to work for sick-listed patients.

The challenges for health personnel is not cure of the patients back pain, but to build up rehabilitation programs which focus on disability and work incapacity, in patients which are at risk of loosing their work. Dr. P. Loisel, Montreal, Canada", has since 1995 treated patients with back pain according to the "The PREVICAP model - (PREVention of work handICAP)", where the main purpose with work-related program is to prevent prolonged disability and to help patients back to work. Loisel demonstrated that the PREVICAP models accelerated the "return to work" factor by a factor 2.4 (p=0.01). The PREVICAP model have also been evaluated in Amsterdam, by Dr. Anema with the same results.

At the Back Clinic, Ullevål University Hospital we have evaluated several exercise programs with good effect on pain and function, but not on the return to work rate. We are planning to do a randomized controlled trial after the PREVICAP model. All included patients in both groups, will have an clinical examination by specialist in Physical Medicine and Rehabilitation and an exercise program. Patients will be randomized to a work-related rehabilitations program or to usual care by the general practitioner.

Hypothesis Main hypothesis: Sick-listed patients with back pain, who will be randomized to the work-related rehabilitation programs, will return to work faster than patients randomized to usual care by the general practitioner.

Second hypothesis: A cost-benefit analysis will favor the exercise program and work place intervention

DETAILED DESCRIPTION:
Background Low back pain is a usual conditions in the western countries and in Norway 40% of the population report decreased function because of back pain. The disease has great economic consequences, which in 2004 came to 15 billions to disability pension and 1,46 billions to physical treatments.

Severe incidence of back pain, like tumours, infections, fractures and pareses are rare and represent less than 1 % of all cases. The main part is within the category of "non-specific low back pain", which is defined as back pain without specific pathology as known cause.

Based on scientific documentation the back-specialists consider non-specific low back pain as a benign and self-limited condition, while patients expect to get treatment because they experience the condition as painful and disabling.

There are several treatments available for patients with "non-specific low back pain". According to the European guidelines exercise and cognitive intervention has good effects on pain and function (www.backpaineurope.org), but it is not documented effect on return to work. In addition it is not documented that treatments which focus on a single treatment neither is effective regarding return to work for sick-listed patients.

It is a usual myth that physical hard work cause back pain. However, only few studies have demonstrated correlations between hard work and sick-leave. On the contrary several studies have demonstrated that back pain is a multifactorial problem, which is not only due to workers' characteristics, but is also closely related to environmental factors, such as the workplace, the healthcare system, the compensation system and the interaction between all stakeholders in the disability problem.

The challenges for health personnel is not cure of the patients back pain, but to build up rehabilitation programs which focus on disability and work incapacity in patients which are at risk of loosing their work.

Dr. P. Loisel, Montreal, Canada", has since 1995 treated patients with back pain according to the "The PREVICAP model - (PREVention of work handICAP)". The main purpose with work-related program is to prevent prolonged disability and to help patients back to work. This approach includes two steps: first identification of factors on the workplace which contribute to the absence of work and second "workplace intervention". Identification of factors at workplace includes physical, ergonomic, psychosocial, interpersonal conflicts and administrative problems. "Workplace intervention" is a rehabilitation program centred at the workplace, allowing a graded transition from the clinical setting to the workplace. Parallel with the workplace intervention the patients enter an exercise-program, adjusted to the workplace intervention.

The PREVICAP models have been evaluated in randomized controlled trials and has accelerated return to work by a factor 2.4 (p=0.01). The most important effect came from the workplace intervention, which alone accelerated the return to work with a factor 1.9 (p=0.01). Patients randomized to the PREVICAP model had 60 days absence from work, compared to 120 days in the control group.

The PREVICAP model have been evaluated in Amsterdam, by Dr. Anema and he demonstrated a significant difference in the return to work rate between patients randomized to "Workplace intervention" and patients randomized to usual treatment.

At the Back Clinic, Ullevål University Hospital we have evaluated several exercise-programs with good effect on pain and function, but not on the return to work rate. This raises an important question: will the return to work rate increase by including workplace intervention to the exercise program and it is possible to implement the PREVICAP model in Norway with the same good results, despite differences between Canada, The Netherlands and Norway with regard to culture, soc-economic conditions, working conditions and compensatory systems.

We are planning to do a randomized controlled trial after the PREVICAP model, where patients sick-listed for back pain will be randomized to either a workplace intervention plus an exercise-program or to an exercise-program alone.

Purpose

The purpose of the project is to answer the following questions:

1. Will more patients return to work and will they do it faster, when they will be included in a work-related rehabilitations program than patients randomized to usual care by the general practitioner, at the follow-up 6 weeks, 3 months, 6 months, 1 and 2 years.
2. Was there significant difference in pain and function between the two groups at the follow-up?
3. Which factors predict the return to work; medical, socioeconomic or factors at the workplace?
4. At the 2 years follow-up- Had the patients had episodes with back pain and in case, how many, of which duration and were they sick-listed for it or did they stay at work?
5. Is there a favorable cost benefit with the program?

The study is a prospective single-blind randomized study. The patients will be randomized by block-randomisation. The randomization will be carried out at a separate locations concealed from the clinical investigators.

Inclusions criteria: Patients with non-specific low back pain sick listed from 6-8 weeks and who are permanently employed. Non-specific low back pain is defined as a back pain not attributable to a recognizable, known specific pathology.

Exclusions criteria: Patients with infection, tumors, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome or cauda equina syndrome, spinal stenosis or spondylolysis/ listesis, serious somatic disease and/or psychic disease and patients with a poor proficiency in Norwegian.

All patients will have a clinical examination of a specialist and a an exercise program. The patients will be randomized to workplace intervention or a control group. Patients randomized to the workplace intervention will be referred to an occupational ergonomist for work site evaluation and return to work program, which include ergonomic conditions and relations to the employer and colleagues. The occupational task of the ergonomists is to organize contacts and meetings between the employer and the patients and make a schedule for return to work. Patients randomized to the control group will go back to their general practitioner for planning return to work.

Sample size:all together 260 patients in the study.

Ethics The study will follow the ethic directions in the Helsinki Declaration and will not be initiated before approval from the National Committee for Research Ethics in Norway. In addition we will also ask for permission to collect and register the data from the Data Inspectorate in Norway. Only patients giving informed consent will be included and they will be informed that they can withdraw from the study at any time and that this will have no otherwise consequences for their treatment.

Registrations of drop-outs The moment time and the cause of drop-outs will be registered. We will attempt to obtain a clinical examination from drop-outs at the 1-year follow-up.

Data analyses and statistic analyses All data will be anonymous coded and registered electronic i SPSS. They will be unidentified in analyses and presentations.

Parametric analyses will be applied on data, which are normally distributed or else, non-parametric statistic will be used. Survival analyses will be used for investigating difference in reduction sickness leave between the two treatment groups. Multivariate analyses will be used for identifying differences in pain, function and fear of avoidance between the two groups. In addition to analysing the data from the patients who completed the trial, the data from dropouts will be analysed according to the intention-to-treat principle.

Preconditions at the Back Clinic for conduction of the study The Back Clinic, Ullevål University Hospital has collaboration with the Compensation system in Oslo, NAV (Norges Arbeids-og Velferdsetat). The surplus from the Back Clinic will be used to employ an occupational ergonomist. The physiotherapists are employees at the Back Clinic and they have tried out the exercise program. Principal investigator (Anne Keller) is applying for grants for a post doc fellowship.

The Back clinic has a test laboratory with a bicycle for testing submaximal oxygen uptake and inclinometer for measuring range of motion of flexion of the back. We have collaboration with Department of neuroradiology for MRI investigations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific low back pain sick listed from 6-8 weeks and who are permanently employed.

Exclusion Criteria:

* Patients with infection, tumors, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome or cauda equina syndrome, spinal stenosis or spondylolysis/ listesis, serious somatic disease and/or psychic disease and patients with a poor proficiency in Norwegian.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is return to work, measured in number of days patients have been sick listed in both groups. | The duration of the project is estimated to 3 years. The project will start January1st 2008 and the inclusion of patients and the follow-up will be in 2008 and 2009. In 2010 follow-up, statistical analyses, writing and publishing the articles.

SECONDARY OUTCOMES:
The secondary outcome measures are improvement in pain, function, stiffness and fear-avoidance beliefs | The duration of the project is estimated to 3 years. The project will start January 1st 2008 and the inclusion of patients and the follow-up will be in 2008 and 2009. In 2010 follow-up, statistical analyses, writing and publishing the articles.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Keller, Dr.Med.Sc, Principal Investigator — Dep of Physical Medicine and Rehab, Ulleval University Hospital, Oslo, Norway
Locations (1):
- Anne Keller, Oslo, Oslo County, Norway